CLINICAL TRIAL: NCT05262153
Title: Clinical and Biochemical Effect of Smoking on Non-surgical Periodontal Treatment in Periodontitis Grade III Stage C Patients
Brief Title: Effect of Smoking on Periodontal Therapy in Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAG-C-DRP-241018-0569
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Periodontal Diseases; Smoking
Keywords: Periodontitis; Smoking; Periodontal treatment
MeSH Terms: conditions — Periodontal Diseases; Smoking; Periodontitis | interventions — Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontally healthy (No Intervention)
- Periodontitis III-C (Active Comparator): The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-surgically performed scaling and root planing
- Periodontitis III-C Smoking (Active Comparator): The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-surgically performed scaling and root planing

INTERVENTIONS:
Procedure: Non-surgically performed scaling and root planing — Treatment of patients with periodontitis was performed using manual and ultrasonic instruments.
  Arms: Periodontitis III-C; Periodontitis III-C Smoking

SUMMARY:
The present study aimed to assess the effect of smoking on non-surgical periodontal treatment on serum and salivary RANKL, OPG and IL34 levels in periodontitis stage III grade C (P-III-C) patients. 20 periodontally healthy, 20 P-III-C and 20 P-III-C with smoking (P-III-CS) participants were enrolled. At baseline, serum and saliva samples were collected and the whole mouth clinical periodontal parameters were recorded. Periodontitis patients received non-surgical periodontal treatment. Clinical parameters were re-measured and samples were re-collected at 1 and 3 months after treatment. Serum and salivary RANKL, OPG and IL34 levels were analyzed by ELISA. Data were analyzed using appropriate statistical tests.

DETAILED DESCRIPTION:
Periodontal disease is an inflammatory process that can result in tooth loss and also is considered a modifying factor for systemic health. In bone tissue, bone resorption by osteoclasts and bone formation by osteoblasts are repeated continuously. Osteoclasts are multinucleated cells that derive from monocyte-/macrophage-lineage cells and resorb bone. In contrast, osteoblasts mediate osteoclastogenesis by expressing receptor activator of nuclear factor-kappa B ligand (RANKL), which is expressed as a membrane-associated cytokine. Osteoprotegerin (OPG) is a soluble RANKL decoy receptor that is predominantly produced by osteoblasts and which prevents osteoclast formation and osteoclastic bone resorption by inhibiting the RANKL-RANKL receptor interaction. IL-34 shares vital functions of M-CSF, and manages myeloid cell survival, differentiation, and proliferation.

This study is the first controlled clinical study that examines the levels of RANKL, OPG and IL-34 in saliva and serum in smoker and non-smoker periodontitis, and evaluates the situation before and after the treatment. The first hypothesis of this study; in smoker periodontitis group, salivary and serum RANKL, OPG and IL-34 levels will be high, in contrast to the non-smoker periodontitis and periodontal healthy group. The second hypothesis of this study is that after periodontal treatment, saliva and serum RANKL and IL-34 levels will decrease, saliva and serum OPG will increase. Based on these hypotheses, the aim of the study is; to compare the levels of RANKL, OPG and IL-34 in saliva and serum of healthy controls, P-III-C, and P-III-CS subjects and to evaluate the effect of periodontal treatment.

A total of 60 systemically healthy patients; 20 periodontally healthy, 20 P-III-C, 20 P-III-CS were included in this study. The whole mouth clinical periodontal examination included measurement of probing depth (PPD), clinical attachment level (CAL), presence of bleeding on probing (BOP), gingival index (GI), and plaque index (PI) at 6 sites per tooth, except the third molars. The presence and type of the alveolar bone loss were assessed on the digital panoramic radiograph in each participant, which was supplemented with periapical radiographs if necessary.

Periodontal status of each patient was evaluated by a single calibrated periodontists with a manual probe. The diagnosis of periodontitis or periodontally health was determined according to the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions.

Treatment

The recruited periodontitis patients received conventional quadrant scaling and root planning (SRP) under local anesthesia in a total of 4 sessions in two weeks. SRP was performed by the same periodontist using ultrasonic inserts and manual periodontal curettes. Re-evaluations were performed at 1 and 3 months following the completion of the SRP. No periodontal intervention was carried out in the periodontally healthy controls.

Saliva and Serum Sampling A total of 5 mL of unstimulated whole saliva was collected by passive drool method between 9:00 and 10:00 am. The participants were advised to avoid food consumption for three hours before sample collection. The participants were seated upright and saliva was collected over a period of 5 minutes with instructions to pool saliva in the floor of the mouth and passively drool it into a sterile glass beaker. Then saliva samples are immediately transferred to a 2 mL polypropylene tube and stored at -80°C. A total of 5 mL of blood was collected from the antecubital fossa by venepuncture method. Serum was isolated from the blood by centrifuging at 5000 rpm for 10 minutes followed by its rapid transfer to a sterile polypropylene tube and storage at -80°C.

Biomarker Immunoassays Saliva and serum samples were thawed on ice. The saliva samples were centrifuged at 5.000 rpm for 15 minutes at room temperature, and supernatants were immediately used for assays. Serum and salivary samples of RANKL, OPG and IL-34 in were measured by ELISA using commercial kits.

Statistical Analysis All statistical analyses were carried out with the standard statistical software package. For the intra-group comparisons, if the data were not normally disturbed, Friedman test and the Dunn test with the Bonferroni correction were used to analyze the change between baseline and 1 month and 3 months after treatment. For inter-group comparisons, Mann-Whitney U test for normally and non-normally disturbed data. The Spearman's rank correlation test was used to detect the correlations of biochemical parameters with clinical parameters and each others in diseased group before and after treatment. All tests were performed at significance level of P <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. systemically healthy individuals
2. having ≥20 teeth present (except third molars)
3. individuals with periodontally healthy, periodontitis stage III grade C diagnoses
4. Smokers were smoking 10 cigarettes per day more than 5 years while non-smokers were never smoked.

Exclusion Criteria:

1. having any diagnosed medical disorders such as diabetes mellitus, cardiovascular diseases, rheumatoid arthritis, immunological and mucocutaneous diseases
2. usage of antibiotics, non-steroidal anti-inflammatory drugs and immunosuppressive agents within the past 6 months
3. having any non-inflammatory destructive periodontal disease
4. nonsurgical/surgical periodontal therapy received in the past year
5. pregnant/ lactating/ postmenopausal females.

Ages: 24 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Salivary IL-34 (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in salivary IL-34 levels from baseline to 1 month and 3 months after treatment
Salivary OPG (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in salivary OPG levels from baseline to 1 month and 3 months after treatment
Salivary RANKL (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in salivary RANKL levels from baseline to 1 month and 3 months after treatment
Serum IL-34 (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in serum IL-34 levels from baseline to 1 month and 3 months after treatment
Serum OPG (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in serum OPG levels from baseline to 1 month and 3 months after treatment
Serum RANKL (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in serum RANKL levels from baseline to 1 month and 3 months after treatment
Sites initially PD≥5mm | baseline to 1 month and 3 months after treatment
  PD reduction in sites initially PD≥5mm

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Faculty of Dentistry, Department of Periodontology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided